CLINICAL TRIAL: NCT03963050
Title: Molecular and Functional Basis of Successful Aging and Frailty
Brief Title: Successful Aging and Frailty
Acronym: SAFe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Massimo Venturelli, PhD, Research Fellow, Universita di Verona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 27111
Record Dates: First submitted 2019-05-17; First posted 2019-05-24 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Frailty Syndrome; Cognitive Impairment; Sarcopenia
Keywords: Frailty phenotype; Cognitive Impairment; Sarcopenia; Exercise
MeSH Terms: conditions — Frailty; Cognitive Dysfunction; Sarcopenia; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CF (Experimental): 30 participants (randomized in 3 groups) with CF will perform a program of intervention for 1 hour a day, 3 days per week, for 1 year.
  Interventions: Other: Exercise Training; Other: Exercise Training + Cognitive Training; Other: Control
- PF (Experimental): 30 participants (randomized in 3 groups) with PF will perform a program of intervention for 1 hour a day, 3 days per week, for 1 year.
  Interventions: Other: Exercise Training; Other: Exercise Training + Cognitive Training; Other: Control

INTERVENTIONS:
Other: Exercise Training — The ET program will consist of endurance exercises at 70% of maximal Heart Rate and resistance exercises at 85% of 1 repetition maximum.
Other: Exercise Training + Cognitive Training — ET: The intervention program will consist of endurance exercises at 70% of maximal Heart Rate and resistance exercises at 85% of 1 repetition maximum.
  CT: The intervention program will be configured as a cognitive rehabilitation and mainly memory rehabilitation: the participants will be trained in practicing restorative and compensatory mnemonic techniques, such as visual imagery, face-name association, calendar, notes and prompts.
Other: Control — NO changes in lifestyle

SUMMARY:
Frailty is the term commonly utilized to describe the geriatric syndrome that exposes the elderly to increased risk of negative health-related events. The frailty phenotypes (PF: physical or CF: cognitive) have demonstrated to predict the major negative health-related outcomes in the old population and show extensive similarities with sarcopenia (for PF) or dementia (for CF). However, the role of neurophysiological and biological factors contributing to the physical and cognitive frail condition, and in particular in which way mitochondrial dysfunction, as well as the hypertrophic and atrophic pathways assessed by genes expression, metabolomics and microbiota composition are contributing to these frail conditions, are still under debate. Therefore, the aim of this trial will be to make evidence based on the behaviors and the strategies that promote healthy lifestyle and successful human aging.

DETAILED DESCRIPTION:
In the majority of the world, the population is living to a greater age. However, older age is usually associated with elevated risk of several pathologies, as well as age-related organ dysfunctions, which in turn can accelerate functional impairments, disability, or death. To identify this geriatric syndrome the term frailty phenotype has been commonly utilized. In particular, the frailty phenotype can be distinguished in physical frailty (PF) phenotype or cognitive frailty (CF) phenotype.

Despite several groups of researchers tried to develop preventive interventions to counteract the physical and cognitive frail condition of elderly, the success of this task has been tempered by the lack of standardized, and universally agreed protocols. Moreover, the limited knowledge of the neurophysiological, and biological determinants of these conditions has precluded important advances in the research of this domain.

Many factors combine to achieve a successful aging: genetics, health care and healty lifestile. Therefore, the aim of the current trial will be to understand the behaviors and the strategies that promote healthy lifestyle and successful human aging.

Oldest old participants with CF and PF will be selected from the neurorehabilitation unit of the University Hospital of Verona (Italy). Healthy oldest old and young participants will be recruited from the section of Movement Sciences of the University of Verona.

After a first phase of neurophysiological and biological examinations that will involve all the 4 groups, only CF and PF participants will be randomly assigned to an intervention program (physical exercise, physical+cognitive exercise or control). Frail participants assigned to exercise groups will then perform 1 year of intervention, 3 days per week, 1 hour per day. Afterwards, the three groups of intervention will undergo the same neurophysiological and biological examinations of the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* YH: 30 healthy young (20-25 years old) participants. They must be free of any disease.
* OH: 30 healthy oldest old (80-90 years old) participants. They must be free of any neural or physical disease and any severe chronic disease (CODP, Heart Failure) that can compromise exercise.
* PF: 30 oldest old (80-90 years old) participants. They must be characterized by functional deficits (sarcopenia, osteoporosis and muscle weakness) without cognitive impairment. Additionally, participants cannot be affected by any severe chronic disease that compromise exercise.
* CF: 30 oldest old (80-90 years old) participants. They must be characterized by mild cognitive impairment (MCI) and subjective cognitive decline without functional deficits. Additionally, participants cannot be affected by any severe chronic disease that compromise exercise.

Exclusion Criteria YH

* Any medication
* Any disease
* General: pregnancy, addictive or previous addictive behavior defined as the abuse of cannabis, opioids or other drugs, carrier of infectious diseases.
* For TMS: Epilepsy, metallic prosthesis, malignant tumor

Exclusion Criteria OH

* Heart failure, angina, pulmonary disease.
* Cognitive frailty (MCI, Alzheimer) or physical frailty (musculoskeletal diseases)
* General: coagulation disorders, pregnancy, addictive or previous addictive behavior defined as the abuse of cannabis, opioids or other drugs, carrier of infectious diseases, suffering from musculoskeletal diseases, suffering from mental illness, inability to cooperate, subjects suffering from known cardiac conditions (e.g., pacemakers, arrhythmias, and cardiac conduction disturbances) or peripheral neuropathy. Moreover, subjects suffering from diabetes, arthritis and under medication will be scored according to specific criteria.
* Assumption of any anticoagulant medication
* Assumption of antiplatelet medications in high dose (es: acetylsalicylic acid >200mg x day)
* For TMS: Epilepsy, metallic prosthesis, malignant tumor
* For MRI: pacemaker, internal defibrillator or other ferromagnetic implants

Exclusion Criteria PF

* Simultaneous presence of physical frailty and cognitive impairment (CDR=0.5)
* For exercise testing and training: heart failure, angina, pulmonary disease.
* General: coagulation disorders, pregnancy, addictive or previous addictive behavior defined as the abuse of cannabis, opioids or other drugs, carrier of infectious diseases, suffering from musculoskeletal diseases, suffering from mental illness, inability to cooperate, subjects suffering from known cardiac conditions (e.g., pacemakers, arrhythmias, and cardiac conduction disturbances) or peripheral neuropathy. Moreover, subjects suffering from diabetes, arthritis and under medication will be scored according to specific criteria.
* The T-scores for the whole body and PA-projection total spine parameters: According to the World Health Organization (WHO) recommendation, participants will be diagnosed as having osteoporosis when the minimum T-score, measured at any site, will be less than -2.5, osteopenia if T-score between -1 and -2.5 and normal if T-score will be greater than -1 according to the World Health Organization guideline. Diagnosis will be made on basis of lowest T score at any measured site (T score ≥-1 SD = Normal; T score between -1 and -2.5 SD = Low bone mass, and T Score ≤-2.5 SD = Osteoporosis). T-score reference values are provided by the DXA scanner manufacturer.
* Assumption of any anticoagulant medication
* Assumption of antiplatelet medications in high dose (es: acetylsalicylic acid >200mg x day)
* For TMS: Epilepsy, metallic prosthesis, malignant tumor
* For MRI: pacemaker, internal defibrillator or other ferromagnetic implants
* Decline a priori to participate in the intervention Phase 2 of the study
* Cut-off exclusion criteria of PF:

  * Fried's Frailty Phenotype: < 3 positive characteristics
  * Timed-up-and-go test: <10 sec
  * The Multidimensional Prognostic Instrument (MPI): < 0.66 score
  * The GAITRite system: > 0.9 m/s
  * Groningen Frailty Indicator: <4

Exclusion Criteria CF

* Simultaneous presence of physical frailty and cognitive impairment (CDR=0.5)
* For exercise testing and training: heart failure, angina, pulmonary disease.
* General: coagulation disorders, pregnancy, addictive or previous addictive behavior defined as the abuse of cannabis, opioids or other drugs, carrier of infectious diseases, suffering from musculoskeletal diseases, suffering from mental illness, inability to cooperate, subjects suffering from known cardiac conditions (e.g., pacemakers, arrhythmias, and cardiac conduction disturbances) or peripheral neuropathy. Moreover, subjects suffering from diabetes, arthritis and under medication will be scored according to specific criteria.
* The T-scores for the whole body and PA-projection total spine parameters: According to the World Health Organization (WHO) recommendation, participants will be diagnosed as having osteoporosis when the minimum T-score, measured at any site, will be less than -2.5, osteopenia if T-score between -1 and -2.5 and normal if T-score will be greater than -1 according to the World Health Organization guideline. Diagnosis will be made on basis of lowest T score at any measured site (T score ≥-1 SD = Normal; T score between -1 and -2.5 SD = Low bone mass, and T Score ≤-2.5 SD = Osteoporosis). T-score reference values are provided by the DXA scanner manufacturer.
* Assumption of any anticoagulant medication
* Assumption of antiplatelet medications in high dose (es: acetylsalicylic acid >200mg x day)
* For TMS: Epilepsy, metallic prosthesis, malignant tumor
* For MRI: pacemaker, internal defibrillator or other ferromagnetic implants
* Decline a priori to participate in the intervention Phase 2 of the study
* Cut-off exclusion criteria of CF:

  * Mini Mental State (MMSE): cut-off 23.8
  * FCSRT: IFR (immediate free recall) cut off <19.59; ITR (immediate total recall) cut off<35; DFR (delayed free recall) cut off <6.31; DTR (delayed total recall) cut off<11; index of sensitivity of cueing cut off<0.9; Number of intrusions cut off>0
  * Digit Span: cut off 3.75
  * Digit Span Reversal (WAIS): cut off 2.65
  * Rey-Osterrieth Complex Figure Test: cut off copy 28.88 - cut off
  * deferred reproduction 9.47
  * Trial Making Test A(ENB2): cut off >93 sec; TMT B (ENB2): cut off >282 sec; TMT B-A (ENB2): cut off>186 sec
  * Frontal Assessment Battery (FAB): cut off <13.4
  * Phonemic Fluency (ENB2): cut off 3
  * Clock Test: cut off <6.25
  * Time up and Go TUG-COG: cut off >15sec
  * Cognitive Function Instrument (partly for the caregiver): no cut-off
  * Neuropsychiatric Inventory (for the caregiver): cut-off >0
  * Geriatric Depression Scale: cut-off>10

Ages: 80 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression of potential biomarkers (circulating miRNA) | 3 years
  Noncoding RNAs, in particular, microRNAs (miRNAs), are a new regulatory system which plays a pivotal role in skeletal muscle adaptation and repairing.
Structural cerebral cortex adaptations (TMS) | 3 years
  Single-pulse TMS will be used to map the brain area representing the vastus lateralis (VL).
Functional cerebral cortex adaptations (TMS) | 3 years
  Single-pulse TMS will be used to investigate the excitability of the corticospinal system. A double-cone coil will be used to stimulate the leg area of the primary motor cortex (M1).
Modifications in the metabolism of cerebral areas (ASL-MRI) | 3 years
  To assess non-invasively cerebral blood flow (CBF)
Muscle mass alterations (DXA) | 3 years
  Muscle mass will be assessed with DXA
Alveolar profiles | 3 years
  Changes in biogenic volatile organic compound concentrations can be used to mirror metabolic or pathophysiological processes in the whole body

SECONDARY OUTCOMES:
Changes in muscular fiber type | 3 years
  Outcome of the changes in fiber typing on the components of the muscle mechanics in each group and Pre-Post intervention in CF and PF groups will be evaluated.
Changes in neuromuscular control 1 | 3 years
  The force rate of development during a maximum voluntary contraction and a tetanic stimulation will be compared in order to estimate the role of central command flow to the muscle in changing the efficiency of the tension development at the tendon.
Changes in neuromuscular control 2 | 3 years
  The EMG envelope rate of development during a maximum voluntary contraction and a tetanic stimulation will be compared in order to estimate the role of central command flow to the muscle in changing the efficiency of the tension development at the tendon.
Mitochondrial Respiration | 3 years
  Changes in mitochondrial respiration function will be measured to asses the level of mitochondrial dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Venturelli, Ph.D., Principal Investigator — Università degli studi di Verona; Maria Romanelli, Ph.D., Principal Investigator — Università degli studi di Verona; Federico Schena, Ph.D., Study Director — Università degli studi di Verona; Lidia Del Piccolo, Ph.D., Study Director — Università degli studi di Verona
Locations (1):
- University of Verona, Verona, Italy

REFERENCES:
- [Result] Hatse S, Brouwers B, Dalmasso B, Laenen A, Kenis C, Schoffski P, Wildiers H. Circulating MicroRNAs as easy-to-measure aging biomarkers in older breast cancer patients: correlation with chronological age but not with fitness/frailty status. PLoS One. 2014 Oct 21;9(10):e110644. doi: 10.1371/journal.pone.0110644. eCollection 2014. PMID 25333486
- [Result] Tan L, Yu JT, Tan MS, Liu QY, Wang HF, Zhang W, Jiang T, Tan L. Genome-wide serum microRNA expression profiling identifies serum biomarkers for Alzheimer's disease. J Alzheimers Dis. 2014;40(4):1017-27. doi: 10.3233/JAD-132144. PMID 24577456
- [Result] Pfaffl MW. A new mathematical model for relative quantification in real-time RT-PCR. Nucleic Acids Res. 2001 May 1;29(9):e45. doi: 10.1093/nar/29.9.e45. PMID 11328886
- [Result] Mayeux R, Stern Y. Epidemiology of Alzheimer disease. Cold Spring Harb Perspect Med. 2012 Aug 1;2(8):a006239. doi: 10.1101/cshperspect.a006239. PMID 22908189
- [Result] Pedrinolla A, Schena F, Venturelli M. Resilience to Alzheimer's Disease: The Role of Physical Activity. Curr Alzheimer Res. 2017 Apr 3;14(5):546 - 553. doi: 10.2174/1567205014666170111145817. PMID 28078981
- [Result] Popa-Wagner A, Mitran S, Sivanesan S, Chang E, Buga AM. ROS and brain diseases: the good, the bad, and the ugly. Oxid Med Cell Longev. 2013;2013:963520. doi: 10.1155/2013/963520. Epub 2013 Dec 5. PMID 24381719
- [Result] Rusanova I, Diaz-Casado ME, Fernandez-Ortiz M, Aranda-Martinez P, Guerra-Librero A, Garcia-Garcia FJ, Escames G, Manas L, Acuna-Castroviejo D. Analysis of Plasma MicroRNAs as Predictors and Biomarkers of Aging and Frailty in Humans. Oxid Med Cell Longev. 2018 Jul 18;2018:7671850. doi: 10.1155/2018/7671850. eCollection 2018. PMID 30116492
- [Result] Princivalle A, Monasta L, Butturini G, Bassi C, Perbellini L. Pancreatic ductal adenocarcinoma can be detected by analysis of volatile organic compounds (VOCs) in alveolar air. BMC Cancer. 2018 May 4;18(1):529. doi: 10.1186/s12885-018-4452-0. PMID 29728093
- [Result] Alsop DC, Detre JA, Golay X, Gunther M, Hendrikse J, Hernandez-Garcia L, Lu H, MacIntosh BJ, Parkes LM, Smits M, van Osch MJ, Wang DJ, Wong EC, Zaharchuk G. Recommended implementation of arterial spin-labeled perfusion MRI for clinical applications: A consensus of the ISMRM perfusion study group and the European consortium for ASL in dementia. Magn Reson Med. 2015 Jan;73(1):102-16. doi: 10.1002/mrm.25197. Epub 2014 Apr 8. PMID 24715426
- [Result] Buxton RB, Frank LR, Wong EC, Siewert B, Warach S, Edelman RR. A general kinetic model for quantitative perfusion imaging with arterial spin labeling. Magn Reson Med. 1998 Sep;40(3):383-96. doi: 10.1002/mrm.1910400308. PMID 9727941
- [Result] Detre JA, Leigh JS, Williams DS, Koretsky AP. Perfusion imaging. Magn Reson Med. 1992 Jan;23(1):37-45. doi: 10.1002/mrm.1910230106. PMID 1734182
- [Result] Du AT, Jahng GH, Hayasaka S, Kramer JH, Rosen HJ, Gorno-Tempini ML, Rankin KP, Miller BL, Weiner MW, Schuff N. Hypoperfusion in frontotemporal dementia and Alzheimer disease by arterial spin labeling MRI. Neurology. 2006 Oct 10;67(7):1215-20. doi: 10.1212/01.wnl.0000238163.71349.78. PMID 17030755